CLINICAL TRIAL: NCT06463730
Title: Comparison of Activity Intensity, Performance, and User's Experience Between Custom and Non-custom Serious Games Combined With Balance Boards for Persons After Stroke
Brief Title: Comparison Between Custom and Non-custom Serious Games Poststroke
Acronym: SeriousGames
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: URIS202402
Record Dates: First submitted 2024-04-18; First posted 2024-06-18 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Stroke
Keywords: Chronic stroke; Active video games; Balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Self-paced first, non-custom first (Experimental): Order of interventions: self-paced non-custom games, self-paced custom games, game-paced non-custom games, game-paced custom games
  Interventions: Behavioral: Serious games
- Self-paced first, custom first (Experimental): Order of interventions: self-paced custom games, self-paced non-custom games, game-paced custom games, game-paced non-custom games
  Interventions: Behavioral: Serious games
- Game-paced first, non-custom first (Experimental): Order of interventions: game-paced non-custom games, gam-paced custom games, self-paced non-custom games, self-paced custom games
  Interventions: Behavioral: Serious games
- Game-paced first, custom first (Experimental): Order of interventions: game-paced custom games, game-paced non-custom games, self-paced custom games, self-paced non-custom games
  Interventions: Behavioral: Serious games

INTERVENTIONS:
Behavioral: Serious games — Custom games played using the Equio system, non-custom Wii Fit games played using the Nintendo Wii Balance Board

SUMMARY:
Serious games for rehabilitation are delivered through systems that are either customised or non-customised. Custom serious games allow for control of feedback, setting of game speed and difficulty, while non-custom games are less adaptable but provide attractive graphics and sounds. The study compared the activity intensity and user experience of persons after stroke while playing custom and non-custom virtual reality balance games that were both game- and self-paced.

DETAILED DESCRIPTION:
Persons in chronic phase poststroke will play 12 games (6 self- and 6 game-paced games) over two sessions (in randomised order). Within each game-type, custom and non-custom games will be played in random order. All games will be played on a balance board, whereby each pair of a custom and non-custom game will require comparable movement directions of the center of pressure. The custom system will be compared to the non-custom system in terms of number of repetitions, movement amplitude, users' enjoyment, flow state, likeability and perception of exertion.

ELIGIBILITY:
Inclusion Criteria:

* chronic phase (>6 months) after stroke
* ability to walk with supervision or independently with or without walking aid on flat ground or all surfaces
* stable health condition
* ability to follow simple instructions

Exclusion Criteria:

* additional neurological condition
* musculoskeletal impairments that would interfere with execution of the required tasks or completing the questionnaires

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Number of repetitions | On the day of the intervention during each game (anticipated duration: 5 minutes)
  Number of pelvic displacements in medio-lateral direction extracted from video-recording using specialised software
Amplitude | On the day of the intervention during each game (anticipated duration: 5 minutes)
  Amplitude of pelvic displacements in medio-lateral direction extracted from video-recording using specialised software

SECONDARY OUTCOMES:
Users' enjoyment | On the day of the intervention after each game (anticipated: every 5 minutes)
  Assessed using the Modified Physical Activity Enjoyment Scale (scale score expressed as percentage; higher scores mean a better outcome)
Flow state | On the day of the intervention after each game (anticipated: every 5 minutes)
  Assessed using the Flow State Scale for Occupational Tasks (scale score range 14-98; higher scores mean a better outcome)
Likeability | On the day of the intervention after each game (anticipated: every 5 minutes)
  Rated on a scale from 1 (least liked) to 6 (most liked)
Perception of exertion | On the day of the intervention after each game (anticipated: every 5 minutes)
  Assessed using the Borg's Scale (scale score range 6-20; higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Urška Puh, PT, PhD, Principal Investigator — University Rehabilitation Institute, Republic of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No